CLINICAL TRIAL: NCT03092115
Title: Feasibility Testing of a Novel mHealth Intervention to Improve Adherence to Antiretroviral Therapy Among HIV+ Men Who Have Sex With Men (MSM) Youth
Brief Title: Youth mHealth Adherence Intervention for HIV+ YMSM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-012173; K23MH102128 (NIH); P30AI045008 (NIH)
Record Dates: First submitted 2017-03-03; First posted 2017-03-27 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: HIV
Keywords: Men who have sex with men (MSM); mHealth; antiretroviral therapy (ART); native android app
MeSH Terms: conditions — Homosexuality

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HIV medication adherence app (Experimental): Youth in this arm will receive a medication adherence application to help them remember to take their HIV treatment medication (antiretroviral therapy) as a supplement to current HIV standard of care.
  Interventions: Device: HIV medication adherence app

INTERVENTIONS:
Device: HIV medication adherence app — A medication adherence mobile application for HIV+ youth. It is a theory-driven, patient-centered, mobile phone-based intervention targeting medication adherence and engagement in care among HIV+ youth with features including, but not limited to: custom avatar, medication reminders, calendar tracking of medication adherence, and anonymous chat function for social support.

SUMMARY:
This study will help determine feasibility, acceptability, and preliminary efficacy of an app for HIV medication adherence over a 3-month period. Participation is 3 months consisting of two study visits: An initial study visit and a 3 month follow up visit with both visits lasting about 60-90 minutes. The participant must use the study application (app) at least once daily, and at study visits, must complete surveys.

DETAILED DESCRIPTION:
Young men who have sex with men (YMSM) are disproportionately affected by HIV in the US and fewer than half of youth who are prescribed antiretroviral therapy (ART) achieve viral suppression. Yet few interventions have been developed to address adherence in this population with unique developmental/psychosocial needs. Mobile technology, which is constantly consumed by youth, has the potential to deliver interventions that provide support and feedback in real time as youth go about their daily lives.

This pilot study will test a theory-driven, patient-centered, mobile phone-based intervention (mHealth app) targeting medication adherence among HIV+ youth. It is a three-month prospective feasibility trial to test a medication adherence mobile application consisting of two study visits: baseline and 3-month follow up.

Data collection consists of app usage, Computer Assisted Self-Interview (CASI) for participant satisfaction with the app, demographics, and mental health and risk behaviors, as well as medical chart abstraction of disease biomarkers (CD4, viral load) and pharmacy refill data.

ELIGIBILITY:
Inclusion Criteria:

1. Males (sex at birth male) age 14 to 24 years.
2. HIV-positive
3. Owns an Android smart phone
4. Within 1-month of initiating antiretroviral therapy (ART) medication, previously failed ART and about to restart an ART regimen, or currently on ART having trouble with adherence (defined as having a detectable viral load above 200 copies/ml).
5. MSM (men who have sex with men)
6. Receiving care at the Children's Hospital of Philadelphia (CHOP) Adolescent HIV clinic at the time of the study

Exclusion Criteria:

1. Females (sex at birth; not gender)
2. Males age 13 years or younger or 25 years and older.
3. HIV-negative or status unknown
4. Not in care at the CHOP Adolescent HIV clinic at the time of the study.
5. Does not own an Android smart phone (iPhone, Blackberry, etc. phone users)
6. Is already ART adherent (defined as having an undetectable or suppressed, <200 copies/ml, viral load) or is not on or going to be on ART during the study period.

Ages: 14 Years to 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Suppressed viral load at 3-months | 3 months
  Percentage of participants with suppressed HIV viral load (≤ 200 copies/mL) at the 3-month follow-up study visit.

SECONDARY OUTCOMES:
Self-reported medication adherence rates by participants at 3 months | 3 months
  Measure participants' self-reported rate of adherence at 3-month study visit using the AIDS Clinical Trials Group (ACTG) adherence 4-day recall question administered through computer-assisted self-interview (CASI) survey.
Medication adherence measure using prescription refill information | 3 months
  Percentage of participants who refilled their ART medication determined from medical chart abstraction at 3-month study visit.
Self-reported medication adherence rates by participants over 3-months within the medication adherence application | 3 months
  Percentage participants self-reported medication adherence over a 3-month period within the mHealth app where participants recorded yes/no on whether they adhered to their ART daily.
Measure participant satisfaction of the medication adherence application at 3-months | 3 months
  Measure participant satisfaction with the medication adherence application at the 3-month study visit measured by a xx-item questionnaire that includes likert scales and open-ended qualitative questions administered through computer-assisted self-interview (CASI) survey.
Suppressed viral load at 6-months | 6 months
  a. Percentage of participants with suppressed HIV viral load (≤ 200 copies/mL) at 6-months through medical chart abstraction to determine if participants remained virally suppressed or reached viral suppression since 3-months. No study visit for participant at 6-months, medical abstraction conducted by study team as labs are conducted as part of routine HIV care.

CONTACTS AND LOCATIONS:
Overall Officials: Nadia L Dowshen, MD, MSHP, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
individual participant data will not be shared with other researchers. If shared, datasets will be deidentified of participant health information.